CLINICAL TRIAL: NCT02844101
Title: Assess Whether Knowledge by the Children and Adolescents of the Function of the Accelerometer Determines Its Amount of Physical Activity
Brief Title: Assess Whether Knowledge by the Younger of the Function of the Accelerometer Determines Its Amount of Physical Activity
Acronym: ACCELORIX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012_29; 2012-A01647-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-07-13; First posted 2016-07-26 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-blinded group (Other): The non-blinded subjects will be informed that the accelerometer device (GT3X Actigraph accelerometer) is an accelerometer that assessed physical activity levels and patterns
  Interventions: Device: GT3X Actigraph accelerometer.
- blinded group (Other): The blinded subjects will be informed that they will test the reliability of a new device for body posture assessment and these youngsters will not receive any information with regards to physical activity.
  Interventions: Device: GT3X Actigraph accelerometer.

INTERVENTIONS:
Device: GT3X Actigraph accelerometer.

SUMMARY:
Eighty healthy youngsters, aged 10-18 years, will be equally randomized between the blinded and the non-blinded group. The blinded subjects will be informed that we were testing the reliability of a new device for body posture assessment and these youngsters will did not receive any information with regards to physical activity. Conversely, the non-blinded subjects were informed that the device was an accelerometer that assessed physical activity levels and patterns. Participants will be instructed to wear the accelerometer for 4 consecutive days and to keep a non-wear log diary over the 4 day-monitoring. The overall duration and the duration relative to the quality of the physical activity patterns (sedentary, light, moderate, vigorous and moderate to vigorous) were computed for each group during the 4-day monitoring, then compared between the two groups using the Student's t test.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years old adolescent
* normal clinical examination,
* normal nutritional status at baseline defined by a weight / height ratio between - 2 and + 2 DS DS

Exclusion Criteria:

* abnormal ECG
* known chronic disease
* acute infection dating back at least a week.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
physical activity by GT3X Actigraph accelerometer. | during 4 days
  The physical activity measured in counts/day using an GT3X Actigraph accelerometer.
  Participants were instructed to wear the accelerometer for 4 consecutive days and to keep a non-wear log diary over the 4 day-monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gottrand, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vanhelst J, Beghin L, Drumez E, Coopman S, Gottrand F. Awareness of wearing an accelerometer does not affect physical activity in youth. BMC Med Res Methodol. 2017 Jul 11;17(1):99. doi: 10.1186/s12874-017-0378-5. PMID 28693500
- [Derived] Vanhelst J, Vidal F, Drumez E, Beghin L, Baudelet JB, Coopman S, Gottrand F. Comparison and validation of accelerometer wear time and non-wear time algorithms for assessing physical activity levels in children and adolescents. BMC Med Res Methodol. 2019 Apr 2;19(1):72. doi: 10.1186/s12874-019-0712-1. PMID 30940079